CLINICAL TRIAL: NCT02980029
Title: Pharmacodynamic Effects of Fatty Acid Synthase (FASN) Inhibition With TVB-2640 in Resectable Colon Cancer and Other Resectable Cancers; a Window Trial.
Brief Title: TVB 2640 for Resectable Colon Cancer Other Resectable Cancers; a Window Trial.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated by the PRMC for low accrual
Sponsor: Mark Evers (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mark Evers, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCC-16-MULTI-22; MCC-16-GI-98 (Other: UK Markey Cancer Center (former protocol number)); R01CA208343 (NIH)
Record Dates: First submitted 2016-10-12; First posted 2016-12-02 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2024-01

CONDITIONS: Colon Cancer
Keywords: Resectable Tumors
MeSH Terms: conditions — Colonic Neoplasms | interventions — TVB-2640

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TVB-2640 (Experimental): TVB-2640 is a potent and reversible inhibitor of the FASN enzyme.
  Interventions: Drug: TVB-2640
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TVB-2640 — TVB-2640 is a potent and reversible inhibitor of the FASN enzyme. TVB-2640 inhibits the β-ketoacyl reductase (KR) enzymatic activity of the FASN enzyme. TVB-2640 is uncompetitive towards both NADPH and acetoacetyl-CoA in inhibiting KR activity.
  Arms: TVB-2640
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Primary Objective

• To evaluate the pharmacodynamic effects on metabolic endpoints (malonyl carnitine and tripalmitin levels) following short-term treatment with TVB-2640 in patients with resectable cancers

Secondary Objectives

* To determine if short-term treatment with TVB-2640 decreases cancer cell proliferation.
* To examine other biological endpoints and determine if TVB-2640 inhibits cell survival signaling and lipid biogenesis.
* To perform comprehensive metabolomic analysis in tumor tissues to identify metabolic alterations induced by TVB-2640 treatment.
* To correlate FASN levels in tumor with metabolic and biological endpoints to determine if FASN inhibition has more pronounced effects in patients with increased expression.

DETAILED DESCRIPTION:
This study will test the hypothesis that inhibition of FASN activity blocks tumor lipid biosynthesis and alters the cellular metabolism in colon and other resectable cancers.

* The study is a randomized, double-blind, placebo-controlled pharmacodynamic study.
* Potentially eligible patients will be screened in the University of Kentucky Markey Cancer Center clinics. Eligible patients with histologically or cytologically confirmed resectable cancers without any distant metastases will be identified. Upon obtaining informed consent, patients will be enrolled into the study and randomized to TVB-2640 or placebo in a 2:1 fashion. Subjects and clinical investigators will be blinded to treatment group assignment.
* Baseline blood samples will be collected on Day 0 for all patients.
* All enrolled patients will receive the study drug (TVB-2640 or placebo) at a BSA-derived flat dose, orally once daily, starting Day 1. They will receive the study drug for 10-21 days (minimum of 10 days and a maximum of 21 days), i.e. from Day 1 to Day 10-21. The last dose of the study drug will be on the day before the surgical resection.
* For patients in both randomization groups, surgery will be performed anytime during the window of Day 11- Day 22. On the day of surgery, surgical resection specimen and blood samples will be collected.
* All patients will be evaluated and graded for adverse events according to the NCI Common Terminology for Adverse Events (CTCAE), version 4.03.
* Patients will be followed for 4 weeks after the last dose of the study drug to monitor for any drug-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, resectable colon cancer without distant metastases, who are candidates for surgical resection of the tumor.
* Willing and able to provide written informed consent prior to initiation of any study procedures.
* Male or female who is ≥ 18 years of age on day of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 (fully active, able to carry out all pre-disease activities without restriction) or 1 (unable to perform physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
* Adequate bone marrow function as evidenced by:

  1. Hemoglobin ≥ 9 g/dL
  2. ANC count ≥ 1.5 X 109/L
  3. Platelets ≥ 100 X 109/L
* No significant ischemic heart disease or myocardial infarction (MI) within 6 months before the first dose of study drug and currently has adequate cardiac function, as evidenced by a left ventricular ejection fraction (LVEF) of ≥ 50% as assessed by multi-gated acquisition (MUGA) or ultrasound/echocardiography (ECHO); and corrected QT interval (QTc) < 470 msec
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female patients of childbearing potential should be willing to use 2 methods of birth control, be surgically sterile, or abstain from heterosexual activity for the course of the study through 90 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy, or documented to be surgically sterile
* Willing to participate in the study and comply with all study requirements.

Exclusion Criteria:

* Inability to swallow oral medications or impairment of GI function or GI disease that may significantly alter drug absorption (including, but not limited to active inflammatory bowel disease, malabsorption syndrome). Concomitant therapy with antacids and anti-emetics is permissible
* History of risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome). Concomitant use of medications with a low risk of QT/QTc prolongation (including, but not limited to diphenhydramine, famotidine, ondansetron) is permissible.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Having received cancer-directed therapy (chemotherapy, radiotherapy, hormonal therapy, biologic or immunotherapy, etc) or an investigational drug within 4 weeks (6 weeks for mitomycin C and nitrosoureas) or 5 half-lives of that agent (whichever is shorter) before the first dose of study drug.
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the prescreening or screening visit through 90 days after the last dose of trial treatment
* Inoperable on the basis of co-existent medical problems
* History of clinically significant dry eye (xerophthalmia) or other corneal abnormality or, if a contact lens wearer, does not agree to abstain from contact lens use from Day 1 through the last dose of study drug.
* Other concurrent disease (cardiovascular, renal, hepatic, etc.) or laboratory abnormality that, in the investigator's opinion would increase the risk of participating in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
Malonyl carnitine and tripalmitin levels will be measured in the preand post-treatment blood samples using mass spectrometry blood samples using mass spectrometry. | Up to 56 Days

SECONDARY OUTCOMES:
Expression of markers of tumor growth and cell proliferation (Ki67, β-catenin, c-Myc, survivin, p-AKT, etc) in the pre- treatment (where available) and post-treatment tumor samples will be evaluated using IHC | Up to 56 Days
FASN levels in the pre-treatment and post-treatment tumor samples will be evaluated using IHCsamples will be evaluated using IHC. | Up to 56 Days
TIP47 levels in pre-treatment (where available) and post-treatment tumor samples will be evaluated using IHC. | Up to 56 Days
Comprehensive profile of cellular metabolites involved in various pathways (glycolysis, PPP, Krebs cycle, glutaminolysis) will be assessed in the post-treatment tumor samples using mass spectrometry analyses. | Up to 56 Days
Mutation status of tumors will be evaluated by the Clearseq comprehensive cancer panel, which targets over 145 cancerassociated genes, including APC, CTNNB1, TP53, PIK3CA, BRAF and KRAS. | Up to 56 Days
Levels of TVB-2640 will be measured in the post-treatment blood samples using mass spectrometry analysis. | Up to 56 Days
Toxicities will be graded as per NCI-CTCAE v4.03, based on recorded adverse events, physical examinations, and clinical laboratory assessments. | Up to 56 Days

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Evers, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No